CLINICAL TRIAL: NCT02005510
Title: Randomized Trial of In-Home Cervical Cancer Screening in Underscreened Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); University of Texas Southwestern Medical Center (Other); National Cancer Institute (NCI) (NIH); University of California, Davis (Other)
Responsible Party: Principal Investigator, Rachel Winer, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 44731; R01CA168598 (NIH)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; screening; human papillomavirus; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Eligibility is assessed weekly over 2.5 years. Study participants are assigned to the control arm or to the intervention arm. After follow-up is complete, control arm participants are re-assessed for eligibility and re-randomization.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-home HPV Screening (Experimental): Usual care PLUS a mailed in-home high-risk HPV testing kit (accompanied by an invitational letter, research information sheet, and illustrated instructions for using the kit). "Usual care" consists of patient-, provider-, clinic- and systems-level services to promote adherence to Pap screening, including an annual birthday letter with Pap screening reminders, telephone outreach from primary care providers, and automatic alerts in the electronic medical record for overdue women.
  Interventions: Behavioral: Mailed in-home high-risk HPV testing kit; Other: Usual care
- Usual Care (Placebo Comparator): Usual care. "Usual care" consists of patient-, provider-, clinic- and systems-level services to promote adherence to Pap screening, including an annual birthday letter with Pap screening reminders, telephone outreach from primary care providers, and automatic alerts in the electronic medical record for overdue women.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Mailed in-home high-risk HPV testing kit
  Arms: In-home HPV Screening
Other: Usual care

SUMMARY:
The purpose of this trial is to determine whether mailing in-home human papillomavirus (HPV) screening kits is effective in increasing uptake of cervical cancer screening and early detection and treatment of cervical neoplasia in underscreened women.

DETAILED DESCRIPTION:
Over half of all cervical cancers in the U.S. are diagnosed in unscreened or underscreened women. New national guidelines identify increasing screening uptake as the number one priority for reducing cervical cancer-related morbidity and mortality. Innovative screening strategies that eliminate the need for clinic-based screening could be highly effective in improving screening compliance while maintaining high-quality care. We propose a large, pragmatic randomized controlled trial within Group Health (a large integrated health care delivery system in Washington State) to compare effectiveness of two programmatic approaches to increasing cervical cancer screening among overdue women. The first approach (control arm) is usual care at Group Health, which consists of patient- and provider-level services to promote adherence to Pap screening, and the second approach (intervention arm) includes usual care plus a mailed in-home high-risk human papillomavirus (hrHPV) screening kit. We will randomize eligible women to the in-home hrHPV screening arm or the usual care arm. Compared to usual care, we hypothesize that in-home hrHPV screening will enhance early detection and treatment of cervical neoplasia and improve compliance with screening. The trial will provide definitive evidence-based data on the impact of an in-home hrHPV screening program in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 30 to 64 years of age
* Have a primary care provider at Group Health
* Received annual "birthday letter" with Pap screening reminder 5 months earlier
* No Pap test in the past 3.4 years
* Continuously enrolled at Group Health for at least 3.4 years
* No hysterectomy

Exclusion Criteria:

* Currently pregnant
* Language interpreter needed
* On "do not contact list" for research studies

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19851 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Winer, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Winer RL, Lin J, Tiro JA, Miglioretti DL, Beatty T, Gao H, Kimbel K, Thayer C, Buist DSM. Effect of Patient Characteristics on Uptake of Screening Using a Mailed Human Papillomavirus Self-sampling Kit: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2244343. doi: 10.1001/jamanetworkopen.2022.44343. PMID 36449291
- [Derived] Winer RL, Lin J, Tiro JA, Miglioretti DL, Beatty T, Gao H, Kimbel K, Thayer C, Buist DSM. Effect of Mailed Human Papillomavirus Test Kits vs Usual Care Reminders on Cervical Cancer Screening Uptake, Precancer Detection, and Treatment: A Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1914729. doi: 10.1001/jamanetworkopen.2019.14729. PMID 31693128

RESULTS

PARTICIPANT FLOW:
Groups:
- In-home HPV Screening: Usual care PLUS a mailed in-home high-risk HPV testing kit (accompanied by an invitational letter, research information sheet, and illustrated instructions for using the kit). "Usual care" consists of patient-, provider-, clinic- and systems-level services to promote adherence to Pap screening, including an annual birthday letter with Pap screening reminders, telephone outreach from primary care providers, and automatic alerts in the electronic medical record for overdue women.
  Mailed in-home high-risk HPV testing kit
  Usual care
- Usual Care: Usual care. "Usual care" consists of patient-, provider-, clinic- and systems-level services to promote adherence to Pap screening, including an annual birthday letter with Pap screening reminders, telephone outreach from primary care providers, and automatic alerts in the electronic medical record for overdue women.
  Usual care
Period: Randomized (Round 1)
Arm/Group | In-home HPV Screening | Usual Care
Started | 8120 (Excludes 163 determined to be ineligible post-randomization due to delays in data warehouse update.) | 8111 (Excludes 196 determined to be ineligible post-randomization due to delays in data warehouse update.)
Completed | 8120 | 8111
Not Completed | 0 | 0
Period: Rerandomized (Round 2)
Arm/Group | In-home HPV Screening | Usual Care
Started | 1631 (Excludes 10 determined to be ineligible post-randomization due to delays in data warehouse update.) | 1585 (Excludes 5 determined to be ineligible post-randomization due to delays in data warehouse update.)
Completed | 1631 | 1585
Not Completed | 0 | 0
Period: Rerandomized (Round 3)
Arm/Group | In-home HPV Screening | Usual Care
Started | 209 (Excludes 5 determined to be ineligible post-randomization due to delays in data warehouse update.) | 195
Completed | 209 | 195
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are not available for 117 participants in the intervention arm who opted out of electronic medical record review.
Groups:
- Total: Total of all reporting groups
Arm/Group | In-home HPV Screening | Usual Care | Total
Number analyzed (Participants) | 9843 | 9891 | 19734
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9843 | 9891 | 19734
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9843 | 9891 | 19734
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 486 | 8761 | 9247
  Not Hispanic or Latino | 8710 | 480 | 9190
  Unknown or Not Reported | 647 | 650 | 1297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 147 | 145 | 292
  Asian | 893 | 880 | 1773
  Native Hawaiian or Other Pacific Islander | 151 | 139 | 290
  Black or African American | 438 | 431 | 869
  White | 7018 | 7111 | 14129
  More than one race | 285 | 283 | 568
  Unknown or Not Reported | 911 | 902 | 1813
Region of Enrollment [Number; unit: participants]
  United States | 9843 | 9891 | 19734

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Diagnosed With Cervical Epithelial Neoplasia Grade 2 or Worse
Description: Histologic diagnosis of cervical intraepithelial neoplasia grade 2 or worse
Time Frame: Assessed for up to 12 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | In-home HPV Screening | Usual Care
Number analyzed (Participants) | 9960 | 9891
Participants | 12 | 8

2. Primary Outcome: Number of Participants That Received Treatment for Cervical Intraepithelial Neoplasia Grade 2 or Worse
Description: Receipt of treatment for cervical intraepithelial neoplasia grade 2 or worse
Time Frame: Assessed for up to 18 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | In-home HPV Screening | Usual Care
Number analyzed (Participants) | 9960 | 9891
Participants | 12 | 7

3. Secondary Outcome: Number of Participants That Completed Uptake of Cervical Cancer Screening
Description: Uptake of cervical cancer screening is defined as either: [1] receipt of a Pap or co-test; [2] self-sample hrHPV-positive (16/18-negative) OR unsatisfactory AND receipt of follow-up diagnostic testing (Pap or co-test or colposcopy); [3] self-sample HPV16/18-positive; or [4] self-sample hrHPV-negative)
  Using an intent-to-treat approach, we will use log-binomial regression to estimate the relative risk for cervical cancer screening uptake for the in-home HPV screening arm versus the usual care arm.
  We will also use log-binomial regression to estimate the effects of EMR-derived patient characteristics (e.g. age, race/ethnicity, geocoded socioeconomic status, geocoded distance form primary care clinic, insurance type, time since last Pap test, tobacco use, obesity, and Charlson comorbidity score) on cervical cancer screening uptake, stratified subdivided by randomization arm.
Time Frame: Assessed for up to 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | In-home HPV Screening | Usual Care
Number analyzed (Participants) | 9960 | 9891
Participants | 2618 | 1719

4. Secondary Outcome: Number of Participants With an Abnormal Screening Result
Description: Screening result that warrants repeat testing, surveillance, or immediate colposcopy (per current guidelines) before returning to a routine screening schedule
  Using an intent-to-treat approach, we will use log-binomial regression to estimate the relative risk for an abnormal screening result for the in-home HPV screening arm versus the usual care arm.
Time Frame: Assessed for up to 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | In-home HPV Screening | Usual Care
Number analyzed (Participants) | 9960 | 9891
Participants | 225 | 114

5. Secondary Outcome: Experiences and Attitudes Associated With In-home HPV Testing Uptake
Description: Experiences and attitudes will be measured with online surveys. A subset of intervention arm participants who do and do not return the in-home HPV kit will be invited to complete a survey (target n=200). We will examine psychosocial factors (e.g., cervical cancer/HPV knowledge, attitudes toward screening), experiences, and reactions to kits. We will compare responses in women who do versus do not return a mailed HPV kit.
Time Frame: Survey invitation mailed 6 months post-randomization
Population: A subset of intervention arm participants who do and do not return the in-home HPV kit will be invited to complete a survey.
Measure: Count of Participants; unit: Participants
Arm/Group | In-home HPV Screening | Usual Care
Number analyzed (Participants) | 1355 | 0
Participants
  Kit returner and responded | 116 |
  Kit returner and did not respond | 156 |
  Kit non-returner and responded | 119 |
  Kit non-returner and did not respond | 964 |

6. Secondary Outcome: Experiences and Attitudes Associated With Follow-up of Positive In-home HPV Testing Results
Description: Intervention arm participants who return in-home HPV kits and test positive for HPV will be invited to complete an in-depth semi-structured interview (target n=50). We will explore patient perspectives following a positive human papillomavirus (HPV) self-sampling result to describe experiences and information needs for this home-based screening modality.
Time Frame: Interview invitation mailed after all recommended clinical follow-up complete OR study follow-up window complete, up to 12 months post-randomization
Population: Intervention arm participants who return in-home HPV kits and test positive for HPV will be invited to complete an in-depth semi-structured interview.
Measure: Count of Participants; unit: Participants
Arm/Group | In-home HPV Screening | Usual Care
Number analyzed (Participants) | 75 | 0
Participants
  Kit HPV positive and interviewed | 46 |
  Kit HPV positive and not-interviewed | 29 |

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | In-home HPV Screening | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/9960 | 0/9891
Serious Adverse Events (participants affected / at risk) | 0/9960 | 0/9891
Other Adverse Events (participants affected / at risk) | 5/9960 | 0/9891
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-home HPV Screening (N=9960) | Usual Care (N=9891)
Light bleeding (General disorders) | 2 (2) | 0 (0)
Discomfort (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02005510/Prot_SAP_000.pdf